CLINICAL TRIAL: NCT05669417
Title: Randomized Controlled Trial of Magnesium Sulfate Versus Placebo on the Prevention of Atrial Fibrillation Post Cardiac Surgery.
Brief Title: Peri-Operative Magnesium Infusion to Prevent Atrial Fibrillation Evaluated.
Acronym: POMPAE
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Futility after interim analysis
Sponsor: HagaZiekenhuis (Other)
Responsible Party: Principal Investigator, Jeroen Ludikhuize, MD, PhD, MSc, HagaZiekenhuis
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: T-21-118
Record Dates: First submitted 2022-12-08; First posted 2022-12-30 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Atrial Fibrillation New Onset
Keywords: Cardiac surgery
MeSH Terms: interventions — Magnesium Sulfate; Magnesium

STUDY DESIGN:
Intervention Model Description: Double blinded RCT
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Magnesium Sulfate (Active Comparator): Magnesium sulfate is the active compound and will be administered to achieve plasma serum level of magnesium between 1.5 and 2.0 mmol/L according to the study protocol.
  Interventions: Drug: Magnesium sulfate
- Ringers Lactate (Placebo Comparator): Ringers Lactate is the comparator/placebo and will be administered according to the study protocol.
  Interventions: Drug: Magnesium sulfate

INTERVENTIONS:
Drug: Magnesium sulfate — Based on serum levels, bolus and or continuous administration is provided as dictated by study protocol.
  Other Names: magnesium

SUMMARY:
Post-operative atrial fibrillation (POAF) is commonly observed in patients post cardiac surgery without a previous history of atrial fibrillation (AF) or other arrythmias. It's associated with significant postoperative complications including infection, bleeding reoperation, increased hospital length of stay (LOHS) and mortality. Magnesium has been identified as a potentially interesting compound with easy access and low toxicity. Hypomagnesemia has been observed frequently immediately after cardiac surgery. Both reduction of abnormal atomicity of atrial myocardium and prolongation of the atrial refractory period caused by administration of magnesium may prevent AF. The POMPAE trial will analyse the effectiveness of MgSO4 versus placebo (double blind randomized trial) in the prevention of POAF after cardiac surgery.

DETAILED DESCRIPTION:
Post-operative atrial fibrillation (POAF) is commonly observed in patients post cardiac surgery without a previous history of atrial fibrillation (AF) or other arrythmias. (1) Within this population, AF is considered to be multifactorial in origin (2) but associated with significant postoperative complications including infection, bleeding reoperation, increased hospital length of stay (LOHS) and mortality. (3,4) Multiple interventions have been tried before including anti-arrhythmic drugs (amiodaron, verapamil, sotalol) and rate reducing agents like beta-blockers. (5-7) Although encouraging results have been found with different regimes, adaptation in clinical practice has been hampered by toxicity (amiodarone) and therapeutic index. Magnesium has been identified as a potentially interesting compound with easy access and low toxicity; besides, hypomagnesemia has been observed frequently immediately after cardiac surgery. (8,9) Both reduction of abnormal activity of atrial myocardium and prolongation of the atrial refractory period caused by administration of magnesium may prevent AF. (10) Magnesium metabolism has identified that less then 1% of the total magnesium content is intravascular and serum levels don't always correlate with intracellular concentrations. (11) Hypomagnesaemia is associated with increased ventricular tachycardia and atrial fibrillation which is likely caused by a reduction in membrane triphosphate (ATP) activity. This results in reduced membrane stabilization due to a reduction in intracellular potassium compared to extracellular concentrations thus increasing electrical excitability. (12) Also measuring the intracellular concentration is difficult and especially in a routine fashion as loading tests followed by 24 hour urine analysis (13) and energy-dispersive X-ray analysis are not available. (14) Administration of magnesium sulphate does however correlate to higher intracellular magnesium concentration compared to placebo. (14) Several studies in different populations have shown a reduction in arrhythmias post magnesium supplementation. (15) Previous studies suggest that magnesium administration after cardiac surgery is effective in reducing the incidence of AF. (16) However, uncertainty remains regarding optimal dose/blood levels, duration and method of magnesium administration. (17) In a recent study using a protocol for administration of magnesium aiming for blood levels between 1.5 and 2.0 mmol/L an absolute reduction of POAF of 15.1% (OR 0.49, 95% CI 0.27-0.92) was demonstrated. (18) Based on this study, we designed the POMPAE trial (Peri-Operative Magnesium infusion to Prevent Atrial fibrillation Evaluated). The POMPAE trial is a double blinded randomized clinical trial to investigate the efficacy of magnesium supplementation and the reduction of POAF.

ELIGIBILITY:
Inclusion Criteria:

* Elective cardiac surgery (valve surgery and/or CABG)
* 18 years and above
* Mentally competent

Exclusion Criteria:

* History of atrial fibrillation (AF) or atrial flutter.
* Concomitant rhythm associated procedures (MAZE (surgical ablation)/PVI (pulmonary vein isolation)).
* Pre-existing severe renal impairment (eGFR<30 ml/min).
* Pre-existing 3rd degree heart block without pacemaker presence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-08-06 (Actual)

PRIMARY OUTCOMES:
Incidence of new-onset postoperative atrial fibrillation (POAF) | First seven postoperative days
  New-onset POAF over a period of 5 minutes or longer

SECONDARY OUTCOMES:
28-day postoperative atrial fibrillation (POAF) post-surgery | 28 days post surgery
  The incidence of POAF in the first 28 days post surgery diagnosed with ECG
Duration of POAF and peak heart rate recorded | 28 days post surgery
  The duration of POAF as recorded in the patient chart including the peak heart rate (in bpm)
Length of hospital stay | Total duration of hospital stay
  The total length of hospital stay from day of admission until hospital discharge irrespective of outcome (diseased, home, rehab etc)
Length of ICU stay | Total length of ICU stay after surgery
  The total length of ICU stay from the moment post surgery until discharge to the ward. Possible readmissions are not part of this outcome parameter
Duration of mechanical ventilation | Total length of mechanical ventilation during ICU stay after surgery
  The total length of invasive mechanical ventilation from the moment post surgery until discharge to the ward. Possible readmissions are not part of this outcome parameter
Duration of inotropic and/or vasopressor support | Total length of inotropic/vasopressor support from induction of anaesthesia until ICU discharge
  The duration of inotropic and/or vasopressor support from the start of anaesthesia until discharge to the ward. Possible readmissions are not part of this outcome parameter
Combined outcome including 28-day post-surgery mortality, stroke, pulmonary embolism, delirium (requiring any form of anti-psychotic medication and/or infection requiring antibiotics | 28 days post surgery
  The incidence of the combined outcome of 28-day mortality (outcome 2), the incidence of stroke as per advise neurology department, pulmonary embolism (Ct diagnosis), delirium requiring antipsychotics and/or the use of antibiotics apart from surgical/ICU prophylaxis.

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Ludikhuize, MD, PhD, Principal Investigator — Medical specialist
Locations (1):
- HagaZiekenhuis, The Hague, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
If required and request is made, this will be discussed within the study group and shared if no concerns are raised.
Supporting Information: Study Protocol, SAP
Time Frame: 2023/2024, a study protocol will be prepared as a separate manuscript and submitted for publication in a peer reviewed journal. This will also include the Statistical Analysis Plan.
Access Criteria: Upon acceptance of the study protocol in a peer reviewed journal, the materials are available online.

REFERENCES:
- [Derived] Meerman M, Buijser M, van den Berg L, van den Heuvel AM, Hoohenkerk G, van Driel V, Munsterman L, de Vroege R, Bailey M, Bellomo R, Ludikhuize J. Magnesium sulphate to prevent perioperative atrial fibrillation in cardiac surgery: a randomized clinical trial : A protocol description of the PeriOperative Magnesium Infusion to Prevent Atrial fibrillation Evaluated (POMPAE) trial. Trials. 2024 Aug 15;25(1):540. doi: 10.1186/s13063-024-08368-3. PMID 39148128